CLINICAL TRIAL: NCT03351751
Title: A PHASE 1, DOUBLE-BLIND (3RD PARTY OPEN), RANDOMIZED, PLACEBO-CONTROLLED, DOSE ESCALATION STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF REPEAT ORAL DOSES OF PF-06372865 IN HEALTHY ADULT SUBJECTS
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Repeat Doses of PF-06372865 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: B7431011
Record Dates: First submitted 2017-10-13; First posted 2017-11-24 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: PF-06372865; Safety; Tolerability; Pharmacokinetics; Multiple dose; Healthy subjects
MeSH Terms: interventions — PF-06372865

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects receiving placebo
  Interventions: Drug: Placebo
- PF-06372865 (Experimental): Subjects receiving PF-06372865
  Interventions: Drug: PF-06372865

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06372865 — PF-06372865
  Arms: PF-06372865

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple repeat oral doses of PF-06372865 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non-childbearing potential and/or male subjects between the ages of 18 and 55 years
2. Body mass index of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
3. Subjects who are willing and able to comply with all study procedures (including being able to swallow up to 8 tablets/dose or 16 tablets/day)
4. For optional Japanese subjects only: Japanese subjects currently residing in the United States who have 4 biologic Japanese grandparents born in Japan

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
2. Subjects with history of sleep apnea
3. Any condition possibly affecting drug absorption (eg, gastrectomy)
4. Positive urine drug test
5. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males
6. Treatment with an investigational drug within 30 days or 5 half-lives of the first dose of PF-06372865 (whichever is longer)
7. Clinically significant orthostatic hypotension at screening or screening supine BP >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), following at least 5 minutes of supine rest
8. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec
9. Subjects with any of the following abnormalities in clinical laboratory tests at screening: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >=1.5x upper limit of normal (ULN); total bilirubin level >=1.5x ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <=ULN
10. Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 60 days after the last dose of PF-06372865
11. Male subjects whose partners are currently pregnant
12. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of PF-06372865
13. Use of herbal supplements or hormone replacement therapy within 28 days prior to the first dose of PF-06372865
14. Blood donation of approximately 1 pint (500 mL) or more within 60 days prior to dosing
15. History of sensitivity to heparin or heparin-induced thrombocytopenia
16. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody
17. Other acute or chronic medical or psychiatric condition including recent or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or PF-06372865 administration or may interfere with the interpretation of study results
18. Subjects with active suicidal ideations or suicidal behavior within 5 years prior to screening
19. Subjects with history of cyclic neutropenia.
20. Subjects with known history of hypersensitivity to benzodiazepines, or for whom benzodiazepines would be contraindicated
21. Subjects who have previously been exposed to, or participated in a study with, PF-06372865
22. Subjects with folate deficiency
23. Subjects who have had an X-ray within 4 weeks prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 28-35 days after last dose of study medication
  Treatment-related AEs are any untoward medical occurrences attributed to study drug in a participant who received study drug. A serious adverse events (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28-35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to study drug is assessed by the investigator. Participants with multiple occurrences of an AE within a category are counted once within the category.
Change From Baseline in Vital Signs | 0, 1, 2, 4, 8, and 12 hours post-dose on Days 1 and 21; also 0 and 2 hours post-dose on Days 4, 8, 11, 14, and 17
  Measurement of systolic and diastolic blood pressure and pulse rate
Change From Baseline in Electrocardiogram (ECG) Parameters | 0, 1, 2, 4, 8, and 12 hours post-dose on Days 1 and 21; also 0 and 2 hours post-dose on Days 4, 8, 11, 14, and 17
  Measurement of the following ECG parameters: QT interval, QTcF, PR interval, RR interval, QRS interval, and heart rate.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to 7-10 days after last dose of study medication
  Lab tests include: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein, folate); urinalysis (decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy); other (follicle stimulating hormone, urine drug screening, hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, human immunodeficiency virus).
Maximum Observed Plasma Concentration (Cmax) for PF-06372865 on Day 1 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Maximum observed plasma concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06372865 on Day 1 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Time to reach maximum observed plasma concentration
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for PF-06372865 on Day 1 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Area under the concentration curve from time 0 to end of the dosing interval. The dosing interval is 12 hours.
Maximum Observed Plasma Concentration (Cmax) for PF-06372865 on Day 21 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Maximum observed plasma concentration
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06372865 on Day 21 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Time to reach maximum observed plasma concentration
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for PF-06372865 on Day 21 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, and 12 hours post-dose
  Area under the concentration curve from time 0 to end of the dosing interval. The dosing interval is 12 hours.
Plasma Half-Life (t1/2) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Day 21
  Time for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431011&StudyName=Gaba+Mad+%2B+Micronucleus
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431011&StudyName=A+Phase+1%2C+Double-blind+%283rd+Party+Open%29%2C+Randomized%2C+Placebo-controlled%2C+Dose+Escalation+Study+To+Investigate+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Repeat+Oral+Doses+Of+Pf-06372865+In+Healthy+Adult+Subjects